CLINICAL TRIAL: NCT00240942
Title: Letrozole in the Treatment of Severe and Recurrent Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345ADE04
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Severe and Recurrent Endometriosis
Keywords: Endometriosis; GnRH analog; Aromataseinhibitor; Letrozole
MeSH Terms: conditions — Endometriosis | interventions — Letrozole

INTERVENTIONS:
Drug: Letrozole

SUMMARY:
Endometriosis is a condition in which abnormal growth of tissue histologically resembling the lining of the uterus (endometrium) is present outside of the uterus. This study will investigate the effect of a daily dose of letrozole compared to GnRH is safe and in addition effective in reducing measurable endometriosis lesions and in reducing pain in patients with active endometriosis which were pretreated with GnRH analogs for 2 months.

ELIGIBILITY:
Inclusion Criteria

* Premenopausal women > 18 years of age.
* Laparoscopic and Histologically confirmed diagnosis of moderate or severe endometriosis according rASRM-Score III and IV
* BMI less than 40 kg/m².
* Patient is sexually abstinent or using mechanical (condoms, diaphragms) or sterilization methods of contraception and is willing to continue using them throughout the study.
* Patient is willing and able to comply with study requirements.
* Written informed consent.

Exclusion Criteria

* Endometriosis stage I-II acc. according to rASRM
* Women with other causes of chronic pelvic pain including infectious, gastrointestinal, musculoskeletal, neurologic or psychiatric.
* Significant abnormalities in the physical or laboratory examination including renal and liver function more than twice the normal range.
* Patient desires pregnancy for the duration of the study, is pregnant or breast feeding.
* GnRH therapy during the last 6 months
* Use of hormonal contraception, selective estrogen receptor modulators, progestins, estrogens, steroids, or ovulation induction in the 4 weeks prior to inclusion into the study.
* Untreated abnormal pap smear or other gynecologic condition.
* History of venous thrombosis events including deep vein thrombosis, pulmonary embolism, or retinal vein thrombosis.
* History of stroke, complicated migraine, or documented transient ischemic attack.
* Known hypersensitivity to any ingredient of the study medication.
* Treatment with other aromatase inhibitors
* Other investigational drugs within the past 30 days and the concomitant use of investigational drugs.
* History of non-compliance to medical regimens, and patients who are considered potentially unreliable.

Additional protocol-defined inclusion / exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Response rates (CR, PR, NC, PD) during treatment of advanced endometrial cancer assessed by tumor marker assessments and radiologic imaging at week 12 then q 12 weeks x 1 year then q 16 weeks

SECONDARY OUTCOMES:
Duration of clinical response
Time to progression of the disease
Correlation of tumour response with pretreatment ER/PR status
Histological grade and aromatase levels

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals